CLINICAL TRIAL: NCT02218528
Title: An Exploratory Study of a Plant-based Ingredient for Reducing the Post-prandial Blood Glucose Response in Healthy Indian Adults, When Administered With a Meal
Brief Title: Effect of a Plant-based Ingredient on Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FDS-NAA-1716
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Starchy meal (Placebo Comparator): No Plant-based ingredient added to a starchy meal
  Interventions: Dietary Supplement: No Plant-based ingredient
- Low dose added to starchy meal (Active Comparator): Plant-based ingredient in low dose added to starchy meal
  Interventions: Dietary Supplement: Plant-based ingredient
- Starchy meal and side dish (Placebo Comparator): No Plant-based ingredient added to starchy meal and side dish
  Interventions: Dietary Supplement: No Plant-based ingredient
- Low dose added to starchy meal and side dish (Active Comparator): Plant-based ingredient in low dose added to starchy meal and side dish
  Interventions: Dietary Supplement: Plant-based ingredient
- Medium dose added to starchy meal and side dish (Active Comparator): Plant-based ingredient in medium dose added to starchy meal and side dish
  Interventions: Dietary Supplement: Plant-based ingredient
- High dose added to starchy meal and side dish (Active Comparator): Plant-based ingredient in high dose added to starchy meal and side dish
  Interventions: Dietary Supplement: Plant-based ingredient

INTERVENTIONS:
Dietary Supplement: Plant-based ingredient
  Arms: High dose added to starchy meal and side dish; Low dose added to starchy meal; Low dose added to starchy meal and side dish; Medium dose added to starchy meal and side dish
Dietary Supplement: No Plant-based ingredient
  Arms: Starchy meal; Starchy meal and side dish

SUMMARY:
The study is designed to determine the extent to which a plant-based ingredient is able to modulate blood glucose response when administered with a meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, age at start of the study ≥ 18 and ≤ 50 years;
* Apparently healthy: no medical conditions which might affect the study measurements, as judged by study physician and/or measured by questionnaire, and/or assessed by haematology, blood chemistry and urinalysis;
* Fasting blood glucose value of subjects is ≥ 3.4 and ≤ 6.1 mmol/litre (i.e. 62-110 mg/dl) at screening;
* Haemoglobin level within clinically acceptable range (for male 12 to 17 gm/dL and for females 11 to 15 gm/dL; both inclusive) as judged by the research physician;
* Body mass index (BMI) ≥ 18,0 and ≤ 25,0 kg/m2;
* Agreeing to be informed about medically relevant personal test-results by study physician;
* Willing to comply to study protocol during study;
* Willing to refrain from drinking of alcohol on and one day before the blood withdrawal;
* Accessible veins on arms as determined by examination at screening;
* Being literate;
* HbA1C ≤ 6.5 % (48 mmol/mol).

Exclusion Criteria:

* Any history of diabetes, hyper- (or hypo-) glycemia or other disorder of glucose metabolism;
* Any history of gastro-intestinal disorders (including frequent diarrhoea for example);
* Blood donation in the past 2 months;
* Reported participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study;
* Reported participation in night shift work two weeks prior to pre-study investigation or during the study. Night work is defined as working between 23.00 PM and 6.00 AM;
* Reported intense sporting activities > 10h/w;
* Consumption of ≥120 ml of alcoholic drinks for males and females in a typical week;
* Drug abuse as indicated by urine analysis;
* Chronic smokers, tobacco chewers and drinkers;
* Use of any medication, including supplements and traditional medicine;
* Reported dietary habits, such as a medically prescribed/slimming diet;
* Not being used to eat breakfast;
* Reported weight loss/gain (>10%) in the last six month before the study;
* Being an employee of Unilever or CRO;
* Allergy or intolerance to food products and aversion to food products provided during the study;
* If female: pregnant or will be planning pregnancy during the study period;
* If female: lactating or has been lactating in the 6 weeks before pre-study investigation and/or during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Positive incremental post-prandial blood glucose area unde the curve | 120 minutes

SECONDARY OUTCOMES:
Positive incremental post-prandial blood glucose area under the curve | 180 minutes
Post-prandial insulin response | 120 minutes
Post-prandial insulin response | 180 minutes
Assessment of gastric emptying rate | 10 hours
  GE50% (time to empty 50% of the gastric content) will be determined with paracetamol

OTHER OUTCOMES:
Cmax | 120 minutes
  peak plasma glucose
Cmax-baseline corrected | 120 minutes
  peak plasma glucose - baseline plasma glucose
Tmax | 120 minutes
  peak time plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ketul Modi, MBBS, Principal Investigator — Lambda Therapeutics Research Ltd (LTRL)
Locations (1):
- Lambda Therapeutics Research Ltd (LTRL), Ahmedabad, India